CLINICAL TRIAL: NCT00917930
Title: Effect of Cardiac Rehabilitation on Glucometabolic State in Non-Diabetic Patients With Chronic Ischemic Heart Disease
Brief Title: Evaluation Rehabilitation on Glycometabolic State in Non-Diabetic Coronary Artery Disease (CAD) Patients
Status: Completed | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: giuseppe rosano, IRCCS San Raffaele Roma
Other Study IDs: 090505
Record Dates: First submitted 2009-06-02; First posted 2009-06-11 (Estimated); Last update posted 2009-06-11 (Estimated); Status verified 2009-06

CONDITIONS: Coronary Artery Disease
Keywords: exercise training; functional recovery; heart diseases; altered glucose metabolism early after an acute cardiac event; non diabetes CAD patients; glycometabolic state
MeSH Terms: conditions — Coronary Artery Disease; Heart Diseases | interventions — Physical Conditioning, Human

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- physical training
  Interventions: Behavioral: physical training

INTERVENTIONS:
Behavioral: physical training — intensive cardiac rehabilitation program

SUMMARY:
The purpose of this study is to evaluate the effects of an intensive Cardiac rehabilitation program on glucose metabolism of non-diabetic coronary artery disease patients.

ELIGIBILITY:
Inclusion Criteria:

* patients admitted to undergo a cycle of in-hospital cardiac rehabilitation
* patients without a previous diagnosis of diabetes mellitus
* patients able to start physical training within three days from admission
* fasting blood glucose at admission < 126 mg/dl

Exclusion Criteria:

* previous diagnosis of diabetes mellitus
* acute coronary events or acute heart failure in the past three months
* physical disabilities that contraindicate training

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: non diabetes patients with coronary artery disease
Sampling Method: Probability Sample
Dates: Start 2006-01; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
to evaluate the effective prevalence of glucose metabolism alterations in patients with chronic ischemic heart disease and stable chronic heart failure, without previous diagnosis of diabetes mellitus

SECONDARY OUTCOMES:
to evaluate the potential beneficial effect of physical training on the glycometabolic state